CLINICAL TRIAL: NCT05803109
Title: Efficacy of Extra Virgin Cold Pressed Coconut Oil With Peppermint Essential Oil as Natural Cleaning Agent for Oral Hygiene Routine on Salivary Streptococcus Mutant Levels Versus The Conventional Oral Hygiene Methods in High Caries Risk Patients: A Randomized Clinical Trial
Brief Title: Efficacy of Coconut Oil With Peppermint Essential for Oral Hygiene Routine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Asmaa Mohamed Reda Ahmed Ali, Assistant lecture, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CairoU 4 7 22
Record Dates: First submitted 2023-01-28; First posted 2023-04-07 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Fluoride Adverse Reaction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Double-blind study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- virgin cold-pressed coconut oil with Peppermint essential oil (Experimental): Patients will be instructed to use one packet of the coco pull healthy blend of organic oil (virgin cold pressed coconut oil with Peppermint essential oil)and swish the oil in the mouth and pull it between teeth for 5 minutes then spit out the oil and brush their teeth with the oil for 2 minutes; such a regimen will be repeated twice daily for three months.
  Interventions: Other: AVIVA-PURE-CocoPull-Organic-made in USA
- The fluoride toothpaste (Colgate Total, (Active Comparator): Patients will be instructed to brush their teeth with the fluoride toothpaste (Colgat Total, 1450 ppm) for 2 minutes; such a regimen will be repeated two times daily for three months and use 10 ml of 0.12% chlorhexidine rinse for 1 min/day, 30 min after tooth brushing before going to bed.
  Interventions: Other: AVIVA-PURE-CocoPull-Organic-made in USA

INTERVENTIONS:
Other: AVIVA-PURE-CocoPull-Organic-made in USA — virgin cold pressed coconut oil with Peppermint essential oil

SUMMARY:
This randomized clinical trial will be conducted to investigate the efficacy of an innovative tooth cleaning agent extra virgin coconut oil with peppermint essential oil by oil pulling and toothbrushing with oil on reducing salivary Streptococcus mutans levels, tooth decay and plaque buildup versus on the counter toothpaste in high caries risk patients.

DETAILED DESCRIPTION:
Everyday use of dental health care products has increased. Therefore, there is a legitimately increased interest of healthcare clinicians and consumers in substances added to the toothpaste with the intention to improve their performance and potential benefits and risks that may arise from it. As there are harmful products in the toothpaste for instance: (Fluoride, Sodium Lauryl Sulphate (SLS), Sodium Saccharin and Triclosan which is assumed that it because local reaction includes oral mucosa irritation and desquamation (stomatitis, glossitis, gingivitis, buccal mucositis), while systemic ones are allergic and acute or chronic toxic reactions. Rational Harmful products in the toothpaste for instance: (Fluoride, Sodium Lauryl Sulphate (SLS), Sodium Saccharin and Triclosan which is assumed that it because local reaction includes oral mucosa irritation and desquamation (stomatitis, glossitis, gingivitis, buccal mucositis), while systemic ones are allergic and acute or chronic toxic reactions.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be recruited in this study, will be medically free.
* Age range 20-50 years
* Patients with high caries risk assessment (0- 30% high caries risk) according to Cariogram - a multifactorial risk assessment model for dental caries.
* Non-Smoking patients
* Not under antibiotic therapy either at the time of the study or up to the last month before the start of the study.
* Male or Female patients
* Patients have brushing habits
* No Fixed orthodontic treatment
* No active or untreated caries
* Patients on non-cariogenic diet

Exclusion Criteria:

* Patients with a compromised medical history.
* Patients with low caries risk assessment according to Cariogram - a multifactorial risk assessment model for dental caries.
* Patients with severe or active periodontal disease.
* Patients with a history of allergy to any of the drugs or chemicals will be used in the study.
* Patients on any antibiotics during the past month.
* Smoking patient
* Patients with very low saliva secretion xerostomia less than 0.5ml stimulated saliva /min score 3 according to Cariogram
* Pregnant female patient
* No brushing habits
* Fixed orthodontic treatment
* Active or untreated caries
* Patients on cariogenic diet

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-08-21 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Change in the actual chance to avoid new lesion will be assessed | T0: Baseline. T1: After one month. T2: After three months
  The Measuring test: Cariogram Model (Karabekiroğlu et al 2017), The Measuring units : Percentage
Change in the bacterial count will be assessed | T0: Baseline. T1: After one month. T2: After three months
  The measuring test:Colony forming unit, The measuring units : Cfu/mm2 (Prabakar et al., 2018)
Change in the salivary pH will be assessed | T0: Baseline. T1: After one month. T2: After three months
  The measuring test: Digital pH meter, The measuring unit : Scoring system, (Sondos et al., 2019) (ordinal)
Change in the Plaque index will be assessed Löe-Silness (Loe 1963) | T0: Baseline. T1: After one month. T2: After three months
  The measuring unit : Plaque index The oral hygiene and plaque amount will be estimated using a mirror and graduated periodontal probe in accordance with Silness and Löe plaque index, which assessed the amount of plaque in the cervical part of the tooth.The Plaque Index System
  * (0) No plaque
  * (1) A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may be seen in situ only after application of disclosing solution or by using the probe on the tooth surface.
  * (2) Moderate accumulation of soft deposit s within the gingival pocket, or the tooth and gingival margin which can be seen with the naked eye.
  * (3) Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
  Löe-Silness (Loe 1963) (Sreenivasan et al.,2016), The Measuring units : Scoring system (ordinal)

SECONDARY OUTCOMES:
Change in the Bacterial virulence will be assessed | T0: Baseline. T1: After one month. T2: After three months
  The Measuring test: Streptococcus mutans acidogenicity by Digital pH meter ,the maximum value is 7.2 less than it is bad value (Bedoya-Correa et al., 2021),the measuring units : Scoring system (ordinal)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry Cairo University, Cairo, Kasr El Ainy, Egypt